CLINICAL TRIAL: NCT07303296
Title: A Dose-ranging Randomized, Open-label Study Evaluating the Effect of Bilateral Intravitreal Injection of GS010 at Two Dose Levels on Visual Acuity and Retinal Mitochondrial Activity in Patients Affected With ND4 Leber Hereditary Optic Neuropathy - The REVISE Study
Brief Title: Efficacy and Safety Study of Bilateral IVT Injection of GS010 at Two Dose Levels in LHON Patients
Acronym: REVISE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GenSight Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-LHON-CLIN-08
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Leber Hereditary Optic Disease
Keywords: Heredity Optic atrophy; leber hereditary optic atrophy; LHON; Eye diseases; gene therapy; AAV2 vectors; Inborn genetic disease; Mitochondrial disease; nervous system disease; Intravitreal injection; neurodegenerative disease; leber disease
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber; Eye Diseases; Genetic Diseases, Inborn; Mitochondrial Diseases; Nervous System Diseases; Neurodegenerative Diseases

STUDY DESIGN:
Intervention Model Description: The objective of the Phase 2 study REVISE is to assess the efficacy, retinal mitochondrial activity and safety of two dose levels (high and low doses) of bilateral GS010 IVT measured by ddPCR in ND4 LHON patients, in order to determine the optimal dose for future development.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GS010 High dose (Active Comparator): GS010, at a dose of 3.9E11 VG/eye (High Dose) in ARM H
  Interventions: Genetic: GS010 High dose
- GS010 Low dose (Active Comparator): GS010, at a dose of 1.3E11 VG/eye (Low Dose) in ARM L.
  Interventions: Genetic: GS010 Low dose

INTERVENTIONS:
Genetic: GS010 High dose — For patients allocated dose H GS010 will be administered at a dose of 3.9E11 VG/eye in a final volume of 90 μL (ARM H).
  Other Names: Lumevoq; GS010; lenadogene nolparvovec
  Arms: GS010 High dose
Genetic: GS010 Low dose — For patients allocated dose L, GS010 will be administered at a dose of 1.3E11 VGVG/eye in a final volume of 30 μL (ARM L).
  Other Names: GS010; Lenadogene nolparvovec; Lumevoq
  Arms: GS010 Low dose

SUMMARY:
The goal of this Clinical trial is to assess the safety and efficacy of GS010 at two dose levels on visual acuity and retinal mitochondrial activity in patients affected with ND4 Leber Hereditary Optic Neuropathy (LHON)

ELIGIBILITY:
Inclusion Criteria:

1. Aged 15 years or older at the time of vision loss onset
2. Clinically manifested vision loss due to ND4 LHON in both eyes
3. BCVA of at least LogMAR +2.39, measured at the FrACT scale, in both eyes
4. Documented results of genotyping showing the presence of pathogenic LHON-associated mutation(s) in the ND4 mitochondrial gene and the absence of other pathogenic LHON-associated mutations in the patient's mitochondrial DNA; absence of pathogenic mutations, other than the ND4 LHON-causing mutation(s), which are known to cause pathology of the optic nerve, retina or afferent visual system. Historic results of genetic analysis are acceptable upon Sponsor approval.
5. Vision loss duration from 6 months to 1.5 years in the first affected eye at the Inclusion visit (Day 1)
6. No limitations to OCT image collection that would prevent high quality, reliable images from being obtained in both eyes, as determined by the reading center
7. Clear ocular media and adequate pupillary dilation to permit thorough ocular examination, as assessed by the Investigator
8. Human immunodeficiency virus (HIV) negative serology
9. Female patients of childbearing potential must agree to use effective methods of birth control for up to 6 months after Treatment visit (Day 0). Male patients must agree to use condoms with their female partners for up to 6 months after Treatment visit (Day 0).
10. Willing and able to comply with the protocol, follow study instructions, attend study visits as required and complete all study assessments
11. Patient - and parent/legal guardian if the patient is under 18 years of age - has provided signed, written informed consent

Exclusion Criteria:

* 1. Any known allergy or hypersensitivity to GS010 or any of its constituents 2. Contraindication to IVT in any eye according to the Investigator's clinical judgment and international guidelines (Avery, 2014) 3. Prior intraocular surgery or procedure or IVT, which occurred 6 months prior to inclusion and is considered of clinical relevance per Investigator assessment, or planned intraocular surgery or procedure 4. Presence of optic neuropathy from any cause except LHON, as determined by the Investigator 5. History of recurrent uveitis (idiopathic or immune-related) or active intraocular inflammation, as determined by the Investigator 6. Indication of a unilateral treatment with GS010, as determined by the Investigator:

  * Unilateral or asymmetric ND4 LHON disease: only one eye affected with a vision loss due to ND4 LHON, and the fellow eye with preserved BCVA (LogMAR 0 or close to 0);
  * Amblyopia: unilateral treatment of the functional eye with a vision loss due to ND4 LHON;
  * Patient's desire for unilateral treatment 7. Ingestion of idebenone less than 7 days prior to the Inclusion visit (Day -1) 8. Inability to tolerate the anti-inflammatory regimen 9. Presence of ocular disease (excluding LHON), or systemic disease, or condition (including medications and laboratory test abnormalities) that could compromise patient safety or interfere with assessment of efficacy and safety, as determined by the Investigator 10. Use of any investigational drug, or device, within 90 days, or 5 half-lives, preceding the Inclusion visit (Day-1), whichever is longer, or plans to participate in another study of an investigational drug or device during the study period 11. Previous treatment with ocular gene therapy in either eye. 12. Pregnancy or breast-feeding

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-05-15 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the BCVA change from baseline to 1.5 years post-treatment in the study eyes. | from baseline to 1.5 years post-treatment

SECONDARY OUTCOMES:
BCVA responder rates from baseline to 1.5 years post-treatment in the study eyes, defined as an improvement of at least -0.2 LogMAR. | from baseline to 1.5 years post-treatment
BCVA change from baseline to 1.5 years post-treatment in both eyes. | from baseline to 1.5 years post-treatment
Difference between ARM H and ARM L in BCVA change from baseline to 1.5 years post-treatment in the study eyes. | from baseline to 1.5 years post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital national des quinze-vingts, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GenSight Biologics website — https://www.gensight-biologics.com/fr/